CLINICAL TRIAL: NCT02214121
Title: Multicenter, Open-label, Randomised, Pharmacokinetic (PK) and Pharmacodynamic (PD) Dose-ranging Phase II Study of Ticagrelor Followed by a Double-blind, Randomised, Parallel-group, Placebo-controlled 4 Weeks Extension Phase in Paediatric Patients With Sickle Cell Disease
Brief Title: A Pharmacokinetic (PK) and Pharmacodynamic (PD) Dose-ranging Phase II Study of Ticagrelor in Paediatric Patients With Sickle Cell Disease
Acronym: HESTIA 1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: D5136C00007; 2014-001006-18 (EudraCT Number)
Record Dates: First submitted 2014-08-08; First posted 2014-08-12 (Estimated); Results first posted 2018-05-11 (Actual); Last update posted 2018-12-14 (Actual); Status verified 2018-11

CONDITIONS: Investigation of Platelet Aggregation in Paediatric Patients With Sickle Cell Disease
Keywords: sickle cell anemia; paediatric
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ticagrelor Dose 1a + Dose 2a (Other): Part A: Ticagrelor Dose 1a and ticagrelor Dose 2a single doses + 1 week repeated dosing Part B: Ticagrelor or placebo 4 weeks repeated dosing.
  Interventions: Drug: Ticagrelor Dose 1a + Dose 2a
- Ticagrelor Dose 1b + Dose 2b (Other): Part A: Ticagrelor Dose 1b and ticagrelor Dose 2b single doses + 1 week repeated dosing. Part B: Ticagrelor or placebo 4 weeks repeated dosing.
  Interventions: Drug: Ticagrelor Dose 1b + Dose 2b

INTERVENTIONS:
Drug: Ticagrelor Dose 1a + Dose 2a — Ticagrelor Dose 1a and ticagrelor Dose 2a single doses + 1 week ticagrelor repeated dosing followed by 4 weeks repeated dosing ticagrelor or placebo.
  Arms: Ticagrelor Dose 1a + Dose 2a
Drug: Ticagrelor Dose 1b + Dose 2b — Ticagrelor Dose 1b and ticagrelor Dose 2b single doses + 1 week ticagrelor repeted dosing followed by 4 weeks repeated dosing ticagrelor or placebo.
  Arms: Ticagrelor Dose 1b + Dose 2b

SUMMARY:
The purpose of this Phase II dose-ranging study is to investigate pharmacokinetic (PK) and pharmacodynamic (PD) properties of various doses of ticagrelor followed by 4 weeks of twice-daily treatment in paediatric patients with sickle cell disease

DETAILED DESCRIPTION:
This is a multicenter, open-label, dose-ranging study of ticagrelor followed by a double blind, placebo-controlled extension phase in paediatric patients with sickle cell disease (SCD).

Part A: Patients will be randomised 1:1 to receive one of two dosing schedules consisting of two single weight-adjusted doses of ticagrelor. Pharmacokinetic (PK) parameters and pharmacodynamic (PD) measurements will be determined following each dose. Platelet aggregation will be measured using the VerifyNow™ P2Y12 assay.

Following these 2 single doses, all patients will receive open-label one-week treatment with ticagrelor twice daily to determine tolerability prior to randomisation into Part B.

Part B: In this part patients will be randomised (2:1 ratio) to ticagrelor twice daily or placebo for a 4-week treatment phase.

During the study, patients will be followed for the occurrence of vaso-occlusive crisis (VOC) and for other disease manifestations such as daily pain, analgesic use and complications of SCD.

ELIGIBILITY:
Inclusion criteria

* Children aged ≥2 to <18 years of age
* Diagnosed with homozygous sickle cell (HbSS) or sickle beta-zero-thalassaemia (HbS/β0)

Exclusion criteria

* At risk for haemorrhagic or bradycardic events
* Significant hepatic impairment
* Renal failure requiring dialysis
* Concomitant oral or intravenous therapy with strong CYP3A4 (cytochrome) inhibitors, CYP3A4 substrates with narrow therapeutic indices, or strong CYP3A4 inducers.
* Surgical procedure planned to occur during the study.
* Patients who are currently pregnant or breastfeeding or planning to become pregnant during the study.
* Patients who have known hypersensitivity or contraindication to ticagrelor.

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 46 (Actual)
Dates: Start 2014-09-11 (Actual); Primary Completion 2017-02-27 (Actual); Study Completion 2017-02-27 (Actual)

CONTACTS AND LOCATIONS:
Locations (16):
- United States (6):
  - Research Site, Orange, California
  - Research Site, Chicago, Illinois
  - Research Site, Detroit, Michigan
  - Research Site, Hershey, Pennsylvania
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Charleston, South Carolina
- Research Site, Toronto, Ontario, Canada
- Kenya (2):
  - Research Site, Kisian
  - Research Site, Nairobi
- Lebanon (2):
  - Research Site, Beirut
  - Research Site, Tripoli
- South Africa (2):
  - Research Site, Parow
  - Research Site, Rondebosch
- United Kingdom (3):
  - Research Site, Cardiff
  - Research Site, London
  - Research Site, Manchester

REFERENCES:
- [Background] Hsu LL, Sarnaik S, Williams S, Amilon C, Wissmar J, Berggren A; HESTIA1 Investigators. A dose-ranging study of ticagrelor in children aged 3-17 years with sickle cell disease: A 2-part phase 2 study. Am J Hematol. 2018 Dec;93(12):1493-1500. doi: 10.1002/ajh.25273. Epub 2018 Oct 2. PMID 30187935
- [Derived] Amilon C, Niazi M, Berggren A, Astrand M, Hamren B. Population Pharmacokinetics/Pharmacodynamics of Ticagrelor in Children with Sickle Cell Disease. Clin Pharmacokinet. 2019 Oct;58(10):1295-1307. doi: 10.1007/s40262-019-00758-0. PMID 30972696

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 24 centres, in 6 countries. The first patient was enrolled to Part A of the study on 11 Sep 2014, and the last patient completed Part B of the study on 27 Feb 2017. Recruitment was stopped due to protocol amendment between 8 September 2015 and 1 June 2016.
Pre-assignment Details: 46 patients were randomised to Part A of the study (open label). Of the patients completing Part A, 25 were randomised to Part B of the study (double blind)
Groups:
- Part A - Ticagrelor: Randomised treatment group for Part A of the study. Relevant for the Part A period.
- Part B - Ticagrelor; Part B - Placebo: Randomised treatment group for Part B of the study. Relevant for the Part B period.
Period: Part A
Arm/Group | Part A - Ticagrelor | Part B - Ticagrelor | Part B - Placebo
Started | 46 | 0 | 0
Completed | 39 | 0 | 0
Not Completed | 7 | 0 | 0
Not completed — Patient decision | 2 | 0 | 0
Not completed — Dev. of study-specific withdrawal crit. | 4 | 0 | 0
Not completed — Other | 1 | 0 | 0
Period: Part B
Arm/Group | Part A - Ticagrelor | Part B - Ticagrelor | Part B - Placebo
Started | 0 | 17 | 8
Completed | 0 | 14 | 7
Not Completed | 0 | 3 | 1
Not completed — Patient decision | 0 | 1 | 0
Not completed — Dev. of study-specific withdrawal crit. | 0 | 2 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: The baseline characteristics are tabulated by the actual treatment group. This differs from the numbers in the Participant Flow since not all randomised patients received IP and one patient receiving treatment not matching the randomised treatment
Groups:
- Part A - Ticagrelor: Actual treatment group for Part A of the study. Relevant for the Part A period.
- Part B - Ticagrelor; Part B - Placebo: Actual treatment group for Part B of the study. Relevant for the Part B period.
- Total: Total of all reporting groups
Arm/Group | Part A - Ticagrelor | Part B - Ticagrelor | Part B - Placebo | Total
Number analyzed (Participants) | 45 | 16 | 7 | 68
Age, Continuous [Mean (Standard Deviation); unit: Years] — Relevant for the Part A period of the study. Population: Including only part A
  Years
    number analyzed (Participants) | 45 | 0 | 0 | 45
    (all) | 11.2 (3.34) |  |  | 11.2 (3.34)
Age, Continuous [Mean (Standard Deviation); unit: Years] — Relevant for the Part B period of the study. Population: Including only part B
  Years
    number analyzed (Participants) | 0 | 16 | 7 | 23
    (all) |  | 10.2 (3.73) | 9.7 (3.35) | 10.0 (3.55)
Sex: Female, Male [Count of Participants; unit: Participants] — Relevant for the Part A period of the study Population: Including only part A
  Participants
    number analyzed (Participants) | 45 | 0 | 0 | 45
    Female | 24 | 0 | 0 | 24
    Male | 21 | 0 | 0 | 21
Sex: Female, Male [Count of Participants; unit: Participants] — Relevant for the Part B period of the study. Population: Including only part B
  Participants
    number analyzed (Participants) | 0 | 16 | 7 | 23
    Female | 0 | 9 | 2 | 11
    Male | 0 | 7 | 5 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Relevant for the Part A period Population: Including only part A
  Participants
    number analyzed (Participants) | 45 | 0 | 0 | 45
    Hispanic or Latino | 1 | 0 | 0 | 1
    Not Hispanic or Latino | 44 | 0 | 0 | 44
    Unknown or Not Reported | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Relevant for the Part B period of the study. Population: Including only part B
  Participants
    number analyzed (Participants) | 0 | 16 | 7 | 23
    Hispanic or Latino | 0 | 1 | 0 | 1
    Not Hispanic or Latino | 0 | 15 | 7 | 22
    Unknown or Not Reported | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Relevant for the Part A period of the study Population: Including only part A
  Participants
    White: number analyzed (Participants) | 45 | 0 | 0 | 45
    White | 10 | 0 | 0 | 10
    Black or African American: number analyzed (Participants) | 45 | 0 | 0 | 45
    Black or African American | 35 | 0 | 0 | 35
    Asian: number analyzed (Participants) | 45 | 0 | 0 | 45
    Asian | 0 | 0 | 0 | 0
    Native Hawaiian or Other Pacific Islander: number analyzed (Participants) | 45 | 0 | 0 | 45
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
    American Indian or Alaska Native: number analyzed (Participants) | 45 | 0 | 0 | 45
    American Indian or Alaska Native | 0 | 0 | 0 | 0
    Other: number analyzed (Participants) | 45 | 0 | 0 | 45
    Other | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Relevant for the Part B period of the study. Population: Including only part B
  Participants
    White: number analyzed (Participants) | 0 | 16 | 7 | 23
    White | 0 | 1 | 0 | 1
    Black or African American: number analyzed (Participants) | 0 | 16 | 7 | 23
    Black or African American | 0 | 15 | 7 | 22
    Asian: number analyzed (Participants) | 0 | 16 | 7 | 23
    Asian | 0 | 0 | 0 | 0
    Native Hawaiian or Other Pacific Islander: number analyzed (Participants) | 0 | 16 | 7 | 23
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
    American Indian or Alaska Native: number analyzed (Participants) | 0 | 16 | 7 | 23
    American Indian or Alaska Native | 0 | 0 | 0 | 0
    Other: number analyzed (Participants) | 0 | 16 | 7 | 23
    Other | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: P2Y12 Reaction Units (PRU) - Part A
Time Frame: PRU measurements are taken in conjunction with single doses at Visit 2 (Day 0) and Visit 3 (Day 7) and after repeated dosing at Visit 4 (Day 14). Up to 8 hours post-dose (6 hours following protocol amendment) Visit 2 and 3, and up to 2 hours Visit 4.
Population: The PD analysis set is a subset of the safety analysis set, including all patients having at least one PRU measured. All patients who received at least one single dose of ticagrelor were included in the safety population (SAF) for Part A. Analysis on the SAF was based on the study medication actually received.
Measure: Mean (Standard Deviation); unit: P2Y12 reaction units
Groups:
- Ticagrelor 0.125 mg/kg; Ticagrelor 0.75 mg/kg: Single dose received at Visit 2.
- Ticagrelor 0.375 mg/kg; Ticagrelor 0.563 mg/kg; Ticagrelor 1.125 mg/kg; Ticagrelor 2.25 mg/kg: Single dose received at Visit 3.
- Ticagrelor 0.125 mg/kg Bid; Ticagrelor 0.563 mg/kg Bid; Ticagrelor 0.75 mg/kg Bid: Repeated bid treatment between Visit 3 and Visit 4.
Arm/Group | Ticagrelor 0.125 mg/kg | Ticagrelor 0.75 mg/kg | Ticagrelor 0.375 mg/kg | Ticagrelor 0.563 mg/kg | Ticagrelor 1.125 mg/kg | Ticagrelor 2.25 mg/kg | Ticagrelor 0.125 mg/kg Bid | Ticagrelor 0.563 mg/kg Bid | Ticagrelor 0.75 mg/kg Bid
Number analyzed (Participants) | 14 | 31 | 7 | 18 | 10 | 9 | 14 | 9 | 17
P2Y12 reaction units
  Pre-dose: number analyzed (Participants) | 14 | 30 | 7 | 17 | 10 | 9 | 1 | 9 | 16
  Pre-dose | 301.6 (46.55) | 268.0 (35.95) | 295.4 (42.30) | 287.7 (34.35) | 283.7 (36.88) | 277.7 (39.36) | 320 (NA) — Mean based on one observation. | 205.4 (53.22) | 214.7 (48.71)
  2 hours post-dose: number analyzed (Participants) | 14 | 31 | 7 | 18 | 10 | 9 | 13 | 9 | 17
  2 hours post-dose | 278.2 (47.20) | 138.4 (70.68) | 229.0 (64.22) | 176.2 (79.53) | 128.9 (37.68) | 79.9 (47.74) | 271.2 (70.35) | 102.0 (72.53) | 152.0 (72.35)
  6 hours post-dose: number analyzed (Participants) | 5 | 28 | 2 | 14 | 9 | 9 | 0 | 0 | 0
  6 hours post-dose | 276.0 (75.43) | 189.0 (69.84) | 266.0 (57.98) | 190.4 (47.78) | 191.2 (57.59) | 141.7 (69.58) |  |  |
  8 hours post-dose: number analyzed (Participants) | 5 | 0 | 3 | 1 | 0 | 0 | 0 | 0 | 0
  8 hours post-dose | 343.0 (38.13) |  | 318.3 (66.43) | 318.0 (NA) — Mean based on one observation. |  |  |  |  |

2. Primary Outcome: P2Y12 Reaction Units (PRU) - Part B
Time Frame: PRU measurements are taken after 4 weeks of double blind treatment at the end of Part B.
Population: The PD analysis set is a subset of the safety analysis set, including all patients having at least one PRU measured. All patients who received at least one dose of randomised study drug, ticagrelor or placebo, will be included in the SAF for Part B. Analysis on the SAF was based on the study medication actually received.
Measure: Mean (Standard Deviation); unit: P2Y12 reaction units
Groups:
- Ticagrelor 0.125 mg/kg Bid; Placebo: Repeated bid treatment during Part B.
Arm/Group | Ticagrelor 0.125 mg/kg Bid | Placebo
Number analyzed (Participants) | 9 | 3
P2Y12 reaction units
  Pre-dose: number analyzed (Participants) | 8 | 3
  Pre-dose | 282.8 (19.26) | 313.3 (20.13)
  2 hours post-dose | 259.6 (61.95) | 217.3 (78.34)

3. Primary Outcome: Maximum Plasma Concentration (Cmax) - Part A
Time Frame: PK measurements (up to 8 hours post-dose) are taken in conjunction with single doses at Visit 2 (Day 0) and Visit 3 (Day 7) and after repeated dosing at Visit 4 (Day 14).
Population: The PK analysis set is a subset of the safety analysis set, including all patients having at least one PK variable calculated. All patients who received at least one single dose of ticagrelor were included in the safety population (SAF) for Part A. Analysis on the SAF was based on the study medication actually received.
Measure: Geometric Mean (Standard Deviation); unit: ng/mL
Arm/Group | Ticagrelor 0.125 mg/kg | Ticagrelor 0.75 mg/kg | Ticagrelor 0.375 mg/kg | Ticagrelor 0.563 mg/kg | Ticagrelor 1.125 mg/kg | Ticagrelor 2.25 mg/kg | Ticagrelor 0.125 mg/kg Bid | Ticagrelor 0.563 mg/kg Bid | Ticagrelor 0.75 mg/kg Bid
Number analyzed (Participants) | 14 | 31 | 7 | 18 | 10 | 9 | 14 | 9 | 17
ng/mL | 15.240 (15.2709) | 162.961 (84.9230) | 52.069 (34.4115) | 96.031 (51.4902) | 269.174 (162.2147) | 566.550 (225.9447) | 13.973 (15.3652) | 111.367 (81.1597) | 157.216 (114.8138)

4. Primary Outcome: Maximum Plasma Concentration (Cmax) - Part B
Time Frame: PK measurements (up to 4 hours post-dose) are taken after 4 weeks of double blind treatment at the end of Part B.
Population: The PK analysis set is a subset of the safety analysis set, including all patients having at least one PK variable calculated. All patients who received at least one dose of randomised study drug, ticagrelor or placebo, will be included in the SAF for Part B. Analysis on the SAF was based on the study medication actually received.
Measure: Geometric Mean (Standard Deviation); unit: ng/mL
Arm/Group | Ticagrelor 0.125 mg/kg Bid
Number analyzed (Participants) | 9
ng/mL | 16.394 (13.3671)

5. Primary Outcome: Area Under the Plasma Concentration Time Curve (AUC) - Part A
Description: The PK parameter presented was derived using a model based analysis and not from a non-compartmental (NCA) analysis.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Geometric Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Ticagrelor 0.125 mg/kg | Ticagrelor 0.75 mg/kg | Ticagrelor 0.375 mg/kg | Ticagrelor 0.563 mg/kg | Ticagrelor 1.125 mg/kg | Ticagrelor 2.25 mg/kg | Ticagrelor 0.125 mg/kg Bid | Ticagrelor 0.563 mg/kg Bid | Ticagrelor 0.75 mg/kg Bid
Number analyzed (Participants) | 14 | 31 | 7 | 18 | 10 | 9 | 14 | 9 | 17
ng*h/mL | 161.9 (72.24) | 1151.9 (308.39) | 437.5 (262.24) | 879.3 (236.12) | 1638.7 (521.80) | 2850.9 (1277.39) | 161.9 (72.24) | 913.5 (208.82) | 1022.4 (287.32)

6. Primary Outcome: Area Under the Plasma Concentration Time Curve (AUC) - Part B
Description: The PK parameter presented was derived using a model based analysis and not from a non-compartmental (NCA) analysis.
Time Frame: PK measurements (up to 4 hours post-dose) are taken after 4 weeks of double blind treatment at the end of Part B.
Population: as for outcome 4
Measure: Geometric Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Ticagrelor 0.125 mg/kg Bid
Number analyzed (Participants) | 9
ng*h/mL | 160.6 (88.58)

7. Secondary Outcome: Assessment of Ticagrelor Concentration - Part A
Time Frame: In conjunction with single doses at Visit 2 (Day 0) and Visit 3 (Day 7), after repeated dosing at Visit 4 (Day 14). Up to 8h post-dose (6h following protocol amendment, no pre-dose) Visit 2 and 3, up to 2h Visit 4 (pre-dose, 1h added following amendment)
Population: as for outcome 3
Measure: Geometric Mean (Standard Deviation); unit: ng/mL
Arm/Group | Ticagrelor 0.125 mg/kg | Ticagrelor 0.75 mg/kg | Ticagrelor 0.375 mg/kg | Ticagrelor 0.563 mg/kg | Ticagrelor 1.125 mg/kg | Ticagrelor 2.25 mg/kg | Ticagrelor 0.125 mg/kg Bid | Ticagrelor 0.563 mg/kg Bid | Ticagrelor 0.75 mg/kg Bid
Number analyzed (Participants) | 14 | 31 | 7 | 18 | 10 | 9 | 14 | 9 | 17
ng/mL
  Pre-dose: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 9 | 16
  Pre-dose |  |  |  |  |  |  | 2.170 (NA) — Mean based on one observation. | 31.937 (48.6501) | 28.066 (27.1344)
  1 hour post-dose: number analyzed (Participants) | 14 | 31 | 7 | 18 | 10 | 9 | 0 | 8 | 17
  1 hour post-dose | 12.713 (16.0627) | 104.243 (103.1502) | 34.069 (42.3746) | 33.294 (55.4258) | 182.558 (188.4254) | 390.568 (294.2189) |  | 80.414 (75.9675) | 151.520 (116.0079)
  2 hours post-dose: number analyzed (Participants) | 14 | 31 | 7 | 18 | 10 | 9 | 14 | 9 | 16
  2 hours post-dose | 11.465 (8.7427) | 107.729 (62.8343) | 37.782 (31.6890) | 74.626 (50.7053) | 162.435 (161.8489) | 426.804 (212.5385) | 13.973 (15.3652) | 102.166 (78.0785) | 101.618 (65.2415)
  4 hours post-dose: number analyzed (Participants) | 14 | 31 | 6 | 18 | 10 | 9 | 0 | 0 | 0
  4 hours post-dose | 6.647 (4.4533) | 75.907 (31.2786) | 20.122 (9.9383) | 51.005 (24.6435) | 118.217 (42.0873) | 188.383 (111.9267) |  |  |
  6 hours post-dose: number analyzed (Participants) | 7 | 31 | 3 | 16 | 10 | 9 | 0 | 0 | 0
  6 hours post-dose | 3.663 (3.4061) | 52.966 (29.0297) | 19.435 (15.7259) | 45.502 (17.8950) | 69.708 (44.3168) | 125.279 (89.0005) |  |  |
  8 hours post-dose: number analyzed (Participants) | 6 | 0 | 3 | 2 | 0 | 0 | 0 | 0 | 0
  8 hours post-dose | 3.880 (3.3171) |  | 15.699 (20.7596) | 15.691 (15.1392) |  |  |  |  |

8. Secondary Outcome: Assessment of Ticagrelor Concentration - Part B
Time Frame: PK measurements (up to 4 hours post-dose) are taken after 4 weeks of double blind treatment at the end of Part B.
Population: as for outcome 3
Measure: Geometric Mean (Standard Deviation); unit: ng/mL
Arm/Group | Ticagrelor 0.125 mg/kg Bid
Number analyzed (Participants) | 9
ng/mL
  Pre-dose: number analyzed (Participants) | 8
  Pre-dose | 2.478 (3.9580)
  1 hour post-dose: number analyzed (Participants) | 7
  1 hour post-dose | 9.677 (9.4275)
  2 hours post-dose | 14.144 (12.4711)
  4 hours post-dose: number analyzed (Participants) | 8
  4 hours post-dose | 9.605 (14.4979)

9. Secondary Outcome: Assessment of AR-C124910XX Concentration - Part A
Description: AR-C124910XX is the active metabolite of Ticagrelor
Time Frame: as for outcome 7
Population: as for outcome 3
Measure: Geometric Mean (Standard Deviation); unit: ng/mL
Arm/Group | Ticagrelor 0.125 mg/kg | Ticagrelor 0.75 mg/kg | Ticagrelor 0.375 mg/kg | Ticagrelor 0.563 mg/kg | Ticagrelor 1.125 mg/kg | Ticagrelor 2.25 mg/kg | Ticagrelor 0.125 mg/kg Bid | Ticagrelor 0.563 mg/kg Bid | Ticagrelor 0.75 mg/kg Bid
Number analyzed (Participants) | 14 | 31 | 7 | 18 | 10 | 9 | 14 | 9 | 17
ng/mL
  Pre-dose: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 9 | 16
  Pre-dose |  |  |  |  |  |  | 1.250 (NA) — Mean based on one observation. | 17.380 (10.0399) | 20.359 (15.0788)
  1 hour post-dose: number analyzed (Participants) | 14 | 31 | 7 | 18 | 10 | 9 | 0 | 8 | 17
  1 hour post-dose | 1.782 (1.6604) | 16.302 (22.4614) | 4.577 (7.8610) | 3.708 (13.3332) | 30.070 (44.2950) | 63.088 (84.2091) |  | 24.945 (15.6547) | 43.986 (29.8127)
  2 hours post-dose: number analyzed (Participants) | 14 | 31 | 7 | 18 | 10 | 9 | 14 | 9 | 16
  2 hours post-dose | 2.681 (2.0733) | 33.256 (25.3854) | 11.757 (13.3322) | 15.918 (17.4849) | 52.932 (69.1056) | 149.772 (71.3624) | 4.026 (4.7624) | 37.013 (32.7650) | 44.690 (31.6577)
  4 hours post-dose: number analyzed (Participants) | 14 | 31 | 6 | 18 | 10 | 9 | 0 | 0 | 0
  4 hours post-dose | 2.071 (1.2770) | 29.860 (13.8726) | 7.630 (6.3730) | 17.015 (7.9272) | 50.887 (25.6964) | 101.370 (44.6207) |  |  |
  6 hours post-dose: number analyzed (Participants) | 7 | 31 | 3 | 16 | 10 | 9 | 0 | 0 | 0
  6 hours post-dose | 1.646 (1.0427) | 25.276 (10.8318) | 9.762 (2.3304) | 16.703 (5.8115) | 35.716 (22.3351) | 76.941 (39.9167) |  |  |
  8 hours post-dose: number analyzed (Participants) | 6 | 0 | 3 | 2 | 0 | 0 | 0 | 0 | 0
  8 hours post-dose | 1.715 (1.0226) |  | 6.176 (6.3168) | 9.232 (2.5385) |  |  |  |  |

10. Secondary Outcome: Assessment of AR-C124910XX Concentration - Part B
Description: AR-C124910XX is the active metabolite of Ticagrelor
Time Frame: PK measurements (up to 4 hours post-dose) are taken after 4 weeks of double blind treatment at the end of Part B.
Population: as for outcome 3
Measure: Geometric Mean (Standard Deviation); unit: ng/mL
Arm/Group | Ticagrelor 0.125 mg/kg Bid
Number analyzed (Participants) | 9
ng/mL
  Pre-dose: number analyzed (Participants) | 8
  Pre-dose | 1.810 (1.1213)
  1 hour post-dose: number analyzed (Participants) | 7
  1 hour post-dose | 2.865 (1.6443)
  2 hours post-dose | 4.160 (3.1503)
  4 hours post-dose: number analyzed (Participants) | 8
  4 hours post-dose | 3.953 (4.1179)

11. Secondary Outcome: Oral Clearance (CL/F) - Part A
Description: The PK parameter presented were derived using a model based analysis and not from a non-compartmental (NCA) analysis.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Geometric Mean (Standard Deviation); unit: L/h
Groups:
- Overall: All patients receiving Ticagrelor during Part A.
Arm/Group | Overall
Number analyzed (Participants) | 45
L/h | 22.50 (7.531)

12. Secondary Outcome: Oral Clearance (CL/F) - Part B
Description: The PK parameter presented was derived using a model based analysis and not from a non-compartmental (NCA) analysis.
Time Frame: PK measurements (up to 4 hours post-dose) are taken after 4 weeks of double blind treatment at the end of Part B.
Population: as for outcome 4
Measure: Geometric Mean (Standard Deviation); unit: L/h
Arm/Group | Ticagrelor 0.125 mg/kg Bid
Number analyzed (Participants) | 9
L/h | 19.15 (6.673)

13. Secondary Outcome: Number of Vaso-occlusive Crises - Part B
Time Frame: During 4 weeks of study treatment starting from randomization in Part B (week 2) up to 4 weeks (week 6).
Population: All patients randomised in Part B were to be included in the efficacy analysis set (EAS). Patients were analysed according to their randomised study medication.
Measure: Mean (Standard Deviation); unit: Number of events
Arm/Group | Part B - Ticagrelor | Part B - Placebo
Number analyzed (Participants) | 15 | 8
Number of events | 1.0 (2.00) | 0.6 (0.74)

14. Secondary Outcome: Number of Vaso-occlusive Crises Requiring Hospitalization or Emergency Department Visits - Part B
Time Frame: During 4 weeks of study treatment starting from randomization in Part B (week 2) up to 4 weeks (week 6).
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: Number of events
Arm/Group | Part B - Ticagrelor | Part B - Placebo
Number analyzed (Participants) | 15 | 8
Number of events | 0.2 (0.41) | 0.1 (0.35)

15. Secondary Outcome: Percentage of Days Hospitalized for Vaso-occlusice Crisis or Other Complications of Sickle Cell Disease - Part B
Time Frame: During 4 weeks of study treatment starting from randomization in Part B (week 2) up to 4 weeks (week 6).
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: Percentage of days
Arm/Group | Part B - Ticagrelor | Part B - Placebo
Number analyzed (Participants) | 15 | 8
Percentage of days | 4.52 (11.816) | 1.34 (3.788)

16. Secondary Outcome: Percentage of Days With Pain (Age >=4) - Part B
Description: Pain measured using the Faces Pain Scale, range 0-10 (0, 2, 4, 6, 8, 10), where 0 is no pain
Time Frame: During 4 weeks of study treatment starting from randomization in Part B (week 2) up to 4 weeks (week 6).
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: Percentage of days
Arm/Group | Part B - Ticagrelor | Part B - Placebo
Number analyzed (Participants) | 14 | 8
Percentage of days | 27.01 (34.065) | 31.78 (23.731)

17. Secondary Outcome: Mean Intensity of Pain (Age >=4) - Part B
Description: Pain measured using the Faces Pain Scale, range 0-10 (0, 2, 4, 6, 8, 10), where 0 is no pain
Time Frame: During 4 weeks of study treatment starting from randomization in Part B (week 2) up to 4 weeks (week 6).
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: Mean score on scale
Arm/Group | Part B - Ticagrelor | Part B - Placebo
Number analyzed (Participants) | 14 | 8
Mean score on scale
  Overall - Part B | 1.40 (2.027) | 0.87 (0.493)
  1st week: number analyzed (Participants) | 13 | 8
  1st week | 1.64 (2.603) | 1.36 (0.827)
  2nd week: number analyzed (Participants) | 13 | 7
  2nd week | 1.11 (2.236) | 0.38 (0.525)
  3rd week: number analyzed (Participants) | 12 | 6
  3rd week | 1.06 (1.881) | 0.67 (1.116)
  4th week: number analyzed (Participants) | 12 | 6
  4th week | 1.46 (2.624) | 0.83 (0.901)

18. Secondary Outcome: Percentage of Days of Analgesic Use (Age >= 4) - Part B
Time Frame: During 4 weeks of study treatment starting from randomization in Part B (week 2) up to 4 weeks (week 6).
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: Percentage of days
Arm/Group | Part B - Ticagrelor | Part B - Placebo
Number analyzed (Participants) | 14 | 8
Percentage of days | 16.79 (20.838) | 18.56 (19.110)

19. Secondary Outcome: Percentage of Days of Opioid Analgesic Use (Age >=4) - Part B
Time Frame: During 4 weeks of study treatment starting from randomization in Part B (week 2) up to 4 weeks (week 6).
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: Percentage of days
Arm/Group | Part B - Ticagrelor | Part B - Placebo
Number analyzed (Participants) | 14 | 8
Percentage of days | 12.46 (22.502) | 0.54 (1.537)

20. Secondary Outcome: Percentage of Days of Absence From School or Work (Age >=6) - Part B
Time Frame: During 4 weeks of study treatment starting from randomization in Part B (week 2) up to 4 weeks (week 6).
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: Percentage of days
Arm/Group | Part B - Ticagrelor | Part B - Placebo
Number analyzed (Participants) | 11 | 6
Percentage of days | 4.87 (10.865) | 5.95 (9.494)

21. Other Pre Specified Outcome: Haemorrhagic Events - Part A
Time Frame: From randomisation to Part A (week 0) through Visit 4 (week 2)
Population: All patients who received at least one single dose of ticagrelor were included in the safety population (SAF) for Part A. Analysis on the SAF was based on the study medication actually received.
Measure: Number; unit: Number of events
Arm/Group | Part A - Ticagrelor
Number analyzed (Participants) | 45
Number of events | 0

22. Other Pre Specified Outcome: Haemorrhagic Events - Part B
Time Frame: During 4 weeks of study treatment starting from randomization in Part B (week 2) up to 4 weeks (week 6).
Population: All patients who received at least one dose of randomised study drug, ticagrelor or placebo, will be included in the SAF for Part B. Analysis on the SAF was based on the study medication actually received. Erroneously treated patients will be accounted for in the actual treatment group.
Measure: Number; unit: Number of events
Arm/Group | Part B - Ticagrelor | Part B - Placebo
Number analyzed (Participants) | 16 | 7
Number of events | 0 | 0

ADVERSE EVENTS:
Time Frame: SAEs were collected from Visit 1 and AEs from Visit 2. SAEs and Other AEs are presented by study period, where Part A consists of the time from randomization to Part A through Visit 4. Part B starts the day after Visit 4 and continues until Visit 8.
Arm/Group | Part A - Ticagrelor | Part B - Ticagrelor | Part B - Placebo
All-Cause Mortality (participants affected / at risk) | 0/45 | 0/16 | 0/7
Serious Adverse Events (participants affected / at risk) | 5/45 | 4/16 | 1/7
Other Adverse Events (participants affected / at risk) | 22/45 | 12/16 | 5/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A - Ticagrelor (N=45) | Part B - Ticagrelor (N=16) | Part B - Placebo (N=7)
Sickle cell anemia with crisis (Blood and lymphatic system disorders) | 3 (3) | 3 (3) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Acute chest syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A - Ticagrelor (N=45) | Part B - Ticagrelor (N=16) | Part B - Placebo (N=7)
Sickle cell anemia with crisis (Blood and lymphatic system disorders) | 6 (8) | 1 (1) | 1 (1)
Tympanic membrane perforation (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 6 (6) | 3 (6) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 3 (3) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 1 (1) | 0 (0)
Facial pain (General disorders) | 2 (4) | 1 (1) | 1 (2)
Non-cardiac chest pain (General disorders) | 2 (2) | 1 (2) | 1 (1)
Pain (General disorders) | 0 (0) | 1 (2) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 2 (2) | 0 (0)
Conjunctivitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Otitis media (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Tinea infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 (7) | 4 (4) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2) | 1 (3)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 (8) | 3 (4) | 2 (2)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 4 (7) | 0 (0) | 2 (2)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
No publication can be made in advance of the first multicenter publication by the sponsor. Any publication will be submitted to the sponsor for review prior to the being published. The sponsor has the right to defer this publication for a period between 60 days to 6 months. The sponsor has the right to restrict the use of confidential information in any of the publications submitted.

DOCUMENTS (2):
  • Statistical Analysis Plan (2017-03-13): https://cdn.clinicaltrials.gov/large-docs/21/NCT02214121/SAP_000.pdf
  • Study Protocol (2015-12-22): https://cdn.clinicaltrials.gov/large-docs/21/NCT02214121/Prot_001.pdf